CLINICAL TRIAL: NCT05178602
Title: The Effect of TaiChi on Ischemic Burden of Patients With Coronary Heart Disease Complicated With Renal Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Ji Huang, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TaiChi trial
Record Dates: First submitted 2021-11-27; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Coronary Heart Disease (CHD); Renal Insufficiency
Keywords: CHD; PCI; Tai Chi; Renal Insufficiency; Cardiac rehabilitation
MeSH Terms: conditions — Coronary Disease; Renal Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): Routine treatment, and tai Chi exercise,5 times a week
  Interventions: Behavioral: Tai Chi Intervention Group
- The control group (No Intervention): Routine treatment, and cardiac rehabilitation is not mandatory

INTERVENTIONS:
Behavioral: Tai Chi Intervention Group — Tai Chi intervention group: routine treatment and tai Chi exercise,5 times a week.
  Arms: The experimental group

SUMMARY:
This study focuses on patients with incomplete revascularization combined with renal insufficiency. And since heart and kidney are two organs influence each other, the study take the mechanism of heart and kidney comorbidity and the risk factors of the two organs.As one of the traditional Chinese sports, Tai Chi is an aerobic exercise combineing movements with static postures, which can significantly improve the aerobic endurance of patients with coronary heart disease. In this study, a parallel, randomized controlled study method is used to quantitatively evaluate the myocardial ischemia condition by myocardial perfusion imaging indicators. This study aims to figure out whether the cardiac rehabilitation training program based on Tai Chi has a positive effect on the patients' myocardial ischemic.

ELIGIBILITY:
Inclusion Criteria:

1. 30-75 years old, all genders;
2. At least two main vessels or their main branch vessels have obvious stenosis (≥50%) according to the coronary angiography;
3. Received stent implantation and incomplete revascularization (incomplete revascularization: at least one vessel whose a diameter> 2.0 mm and at least one lesion with a stenosis> 50%, after PCI);
4. eGFR<60ml/min·1.73m2;
5. Willing to be treated and followed-up during the specified time of the study;
6. Signed the informed consent approved by the Ethics Committee

Exclusion Criteria:

1. Patients with high-risks according to the exercise rehabilitation risks of patients with heart disease by AACVPR;
2. Severe cardiac insufficiency or cardiogenic shock;
3. Combined with severe ventricular arrhythmia, ICD is required;
4. Combined with severe pulmonary hypertension, chronic obstructive pulmonary disease, severe infectious disease, blood system disease, malignant tumor, severe liver damage, etc.;
5. Nervous, mental and motor system diseases;
6. Unwilling to be followed-up.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Nuclein myocardial perfusion Imaging-total scores of stress perfusion（SSS） | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The total load perfusion score indicates the extent and severity of abnormal exercise perfusion. Higher scores indicate more severe myocardial ischemia.
Nuclein myocardial perfusion Imaging-total scores of rest perfusion（SRS） | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The total resting perfusion score (SRS) refers to the degree of myocardial ischemia at rest, with higher scores indicating more severe myocardial ischemia.
Nuclein myocardial perfusion Imaging-Total myocardial ischemia score | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The total myocardial ischemia score reflects the extent and severity of exercise-induced ischemia, with higher scores indicating more severe myocardial ischemia.
Left ventricular ejection fraction difference（△LVEF） | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  ΔLVEF refers to the difference between the subject's post-test ejection fraction and the pre-test ejection fraction, with a larger difference indicating better improvement in cardiac function.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test-Peak oxygen uptake (PVO2) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  Peak oxygen uptake is an important indicator of cardiopulmonary exercise function, it is the golden indicator to assess aerobic exercise capacity, the greater the peak oxygen uptake, the better the cardiopulmonary function. The unit is mL/(min-kg).
Cardiopulmonary exercise test-Oxygen uptake to power ratio（ΔVO2/ΔＷＲ） | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The lower the oxygen uptake to power ratio, the worse the cardiorespiratory function.The unit is mL/(min·W) .
Cardiopulmonary exercise test-Metabolic equivalents (MET) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  Metabolic equivalent is an important indicator in cardiac rehabilitation, which is used to quantify various activities and to determine the intensity of exercise. The higher the metabolic equivalent, the better the cardiopulmonary function.
Cardiopulmonary exercise test-Carbon dioxide ventilation equivalent（VE/VCO2） | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The higher the ratio of VE/VCO2, the lower the ventilation efficiency
Total serum cholesterol(TC) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  Total serum cholesterol level is one of the risk factors for coronary heart disease, and the higher the total serum cholesterol level, the worse it is for cardiovascular.
High-density lipoprotein cholesterol (HDL-C) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The higher the HDL cholesterol in the blood, the better it is for the cardiovascular system.
Low-density lipoprotein cholesterol (LDL-C) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  Low-density lipoprotein cholesterol is one of the risk factors for coronary heart disease, and the higher the Low-density lipoprotein cholesterol level, the worse it is for cardiovascular.
Triglycerides (TG) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  Triglycerides is one of the risk factors for coronary heart disease, and the higher the triglycerides level, the worse it is for cardiovascular.
Body Mass Index(BMI) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The normal value of BMI is between 20kg/m^2 and 25kg/m^2, more than 25kg/m^2 is overweight and more than 30kg/m^2 is obese.
Assess the quality of life | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  In this study, the Seattle Angina Questionnaire (SAQ) was used to measure the quality of life. The higher the patient's score on this questionnaire, the better the quality of life.
Self-rating anxiety scale(SAS) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The higher the score on the self-rating scale of anxiety, the more likely it is that anxiety is present.
Self-Rating Depression scale(SDS) | The intervention lasted for 12 weeks, and the evaluations were carried out before exercise rehabilitation and after the 12-week intervention. All patients were followed up for 1 year, and were reevaluated then.
  The higher the score on the self-rating scale of anxiety, the more likely it is that depression is present.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No